CLINICAL TRIAL: NCT05184244
Title: Investigation of the Psychometric Properties of the Turkish Adaptation of the Activity Limitations in Cerebral Palsy Questionnaire
Brief Title: Turkish Adaptation of the Activity Limitations in Cerebral Palsy Questionnaire
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: IKC444
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Activity, Motor; Cerebral Palsy; Limitation, Mobility
Keywords: cerebral palsy; limitation; activity
MeSH Terms: conditions — Motor Activity; Cerebral Palsy; Mobility Limitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with CP: Children with CP
  Interventions: Other: Activity Limitation Assessment

INTERVENTIONS:
Other: Activity Limitation Assessment — The ACTIVLIM-CP scale evaluates the global activity performance and combined movements of the body.

SUMMARY:
This study aimed to make the Turkish adaptation of ACTIVLIM-CP and to examine its psychometric properties. Eighty-nine individuals with CP, aged between 2-18 years were included in the study. PEDİ, ABILOCO-Kids, and ABILHAND-Kids scores and Wee-FIM questionnaires were used for validity analysis. Test re-test method was used for reliability.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a clinical picture with permanent disorders of the development of movement and posture whether assessing activity limitations matters. This study aimed to make the Turkish adaptation of ACTIVLIM-CP and to examine its psychometric properties.

The internal consistency of the scale was evaluated using Cronbach's alpha value and the inter-measurement reliability using the intraclass correlation coefficient (ICC). In construct validity analysis; ACTIVLIM-CP score; was correlated with PEDİ, ABILOCO-Kids, and ABILHAND-Kids scores and Wee-FIM total scores. A known group comparison was made according to ambulation and epilepsy existence with the Principal Components Explanatory Factor Analysis.

ELIGIBILITY:
Inclusion Criteria:

* children with CP who were diagnosed by a child neurologist
* having physical therapy sessions at special education and rehabilitation center
* age between 2 and 18

Exclusion Criteria:

* whose parent was illiterate or doesn't speak Turkish
* whose parent wasn't complete the questionnaires

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children with CP aged between 2 and 18 years and their parents
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Global Activity Performance assessment | 15 minutes
  ACTIVLIM-CP: Caregiver rates the difficulty degree of 43 activities easy/difficult/impossible/unknown). Questionnaire scores between 0 and 86 points. A higher score shows better activity performance

SECONDARY OUTCOMES:
Gunctional capabilities and limitations | 5 minutes
  Gross Motor Function Classification System: It classifies the motor function of a child from level 1 (slightly affected) to level 5 (severely affected)
Functional independence measurement | 15 minutes
  Functional Independence Measure for Children: The scale includes 18 measurement items and every item scores between 1 -7. A higher score shows more independence
Child's ability to walk assessment | 10 minutes
  Abiloco-Kids: It consists of 10 questions for evaluating the walking performance from the viewpoint of the caregiver. Questionnaire scores between 0 and 20 points. A higher score shows better activity performance
child's manual ability assessment | 15 minutes
  Abilhand-Kids: It consists of 21 questions to measure the manual ability from the viewpoint of the family. Questionnaire scores between 0 and 42 points. A higher score shows better activity performance.
Functional assessment | 20 minutes
  Pediatric Evaluation of Disability Inventory (PEDI): It consists of three Functional Skills Scales, three Caregiver Assistance Scales, and three Modification Scales in the content areas of self-care, mobility, and social function. Functional Skills has 197 items and each item scores as 1(able) and 2(unable), Caregiver Assistance scores between 0(dependent) -5(independent) and Modifications assessing with frequencies .

CONTACTS AND LOCATIONS:
Locations (1):
- İlknur Naz Gürşan, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kinik M, Naz I. An investigation of the psychometric properties of the Turkish adaptation of the activity limitations in cerebral palsy questionnaire. Disabil Rehabil. 2023 Aug;45(16):2668-2674. doi: 10.1080/09638288.2022.2099586. Epub 2022 Jul 22. PMID 35866563